CLINICAL TRIAL: NCT04881825
Title: A 104-Week, Multicenter, Single-Arm, Long-Term, Phase 3 Extension Trial Investigating the Safety and Efficacy of Glepaglutide in Adult Patients With Short Bowel Syndrome (SBS) Completing the EASE SBS 2 Trial
Brief Title: Evaluation of Long Term Safety and Efficacy of Glepaglutide in Treatment of SBS - Extension Trial
Acronym: EASE SBS 3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZP1848-20110; 2020-005502-25 (EudraCT Number); U1111-1261-3358 (Other: WHO)
Record Dates: First submitted 2021-04-22; First posted 2021-05-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- once-weekly glepaglutide (Experimental): All participants will receive 10 mg of glepaglutide as once-weekly injections under the skin (subcutaneous, s.c.)
  Interventions: Drug: Glepaglutide

INTERVENTIONS:
Drug: Glepaglutide — Glepaglutide will be delivered in a single-use autoinjector.
  Other Names: ZP1848

SUMMARY:
This trial is an extension trial to EASE SBS 2. The study looks at whether glepaglutide is a safe treatment for participants with Short Bowel Syndrome (SBS), as well as how well effectiveness is maintained during long term treatment. Participants in this trial will receive glepaglutide as once-weekly injections under the skin (subcutaneous, s.c.) for approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activity
* Completed the full treatment period of the extension trial EASE SBS 2 (ZP1848-17127)

Exclusion Criteria:

* Any condition, disease, or circumstance that in the Investigator's opinion would put the patient at any undue risk, prevent completion of the trial, or confound the planned assessments of the trial
* Not having a colonoscopy performed at End of Trial in EASE SBS 2 (for patients with remnant colon). Note. The results of the colonoscopy must not give rise to any safety concerns. A colonoscopy performed within 6 months prior to End of Trial and not giving rise to any safety concerns is accepted. For patients with a remnant colon, which is not connected to the passage of foods and is thereby dormant, a computerized tomography (CT) scan or magnetic resonance imaging (MRI) will suffice at the discretion of the Investigator
* Use of GLP-1, GLP-2, human growth hormone (HGH), dipeptidyl peptidase-4 (DPP-4) inhibitors, somatostatin, or analogs thereof within 3 months. Note: Prior use of glepaglutide trial drug is allowed
* Females of childbearing potential, who are pregnant, breast-feeding, intend to become pregnant, or are not using highly effective contraceptive methods

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and type of Adverse Events (AEs) | After 108 weeks
  For AEs with onset or worsening following Visit 1

SECONDARY OUTCOMES:
Incidence and type of Serious Adverse Events (SAEs) | After 108 weeks
  For AEs with onset or worsening following Visit 1
Incidence and type of Adverse Events of Special Interest (AESIs) | After 108 weeks
  For AEs with onset or worsening following Visit 1
Change in body temperature | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in heart rate | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in blood pressure | Week 0 in lead-in trial (EASE SBS 1), Week 108
  Seated diastolic and systolic blood pressure
Change in body weight | Week 0 in lead-in trial (EASE SBS 1), Week 108
Number of participants with clinically significant changes in 12-Lead electrocardiogram (ECG) | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in hematology - hemoglobin | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in hematology - hematocrit | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in hematology - white blood cell count | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in hematology - platelet count | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - sodium | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - potassium | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - chloride | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - bicarbonate | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - blood urea nitrogen | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - creatinine | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - creatinine clearance | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - glucose | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - calcium | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - phosphorous | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - alkaline phosphatase | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - alanine aminotransferase (ALT) | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - aspartate aminotransferase (AST) | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - International Normalized Ratio (INR) | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - gamma-glutamyl transferase (GGT) | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - lactic dehydrogenase | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - conjugated bilirubin | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - total bilirubin | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - total protein | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - albumin | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - amylase | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - uric acid | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in biochemistry - C-reactive protein | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in urinalysis - blood | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in urinalysis - glucose | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in urinalysis - leukocytes | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in urinalysis - pH | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in urinalysis - osmolality | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in urinalysis - protein | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in urinalysis - sodium | Week 0 in lead-in trial (EASE SBS 1), Week 108
Change in urinalysis - potassium | Week 0 in lead-in trial (EASE SBS 1), Week 108
Anti-glepaglutide antibodies | Week 0, Week 108
Antibody reactivity to ZP1848 | Week 0, Week 108
Cross-reactivity to glucagon-like peptide-2 (GLP-2) | Week 0, Week 108
Glepaglutide neutralizing antibodies | Week 0, Week 108
Reduction in weekly Parenteral Support (PS) volume | Week 0 in lead-in trial (EASE SBS 1), Week 108
Reduction of at least 20 percent in weekly PS volume | Week 0 in lead-in trial (EASE SBS 1), Week 108
Reduction in days on PS greater than or equal to 1 day per week | Week 0 in lead-in trial (EASE SBS 1), Week 108
Reduction in weekly PS volume of 100 percent (weaned off) | Week 0 in lead-in trial (EASE SBS 1), Week 108

CONTACTS AND LOCATIONS:
Overall Officials: Zealand Pharma, Study Director — Zealand Pharma
Locations (19):
- United States (4):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic College of Medicin, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Vanderbilt University Medical Center, Nashville, Nashville, Tennessee
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Hôpital Beaujon, Clichy
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Frankfurt, Frankfurt
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - Universitätsmedizin Rostock, Rostock
- UMC Radboud Nijmegen, Nijmegen, Netherlands
- Poland (2):
  - Wojewodzki Specjalistyczny Szpital im. M. Pirogowa w Lodzi, Lodz
  - Szpital Skawina sp. z o.o. im. Stanley Dudricka, Skawina
- United Kingdom (3):
  - St Mark's Hospital, Harrow
  - UCLH Foundation NHS Trust, London
  - Norfolk and Norwich University Hospitals, Norwich

IPD SHARING:
Plan to Share IPD: No